CLINICAL TRIAL: NCT02145455
Title: Unity Total Knee Replacement: Prospective Single-centre Clinical Study
Brief Title: Unity Total Knee Replacement Using Two Different Surgical Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSP2013-08
Record Dates: First submitted 2014-05-20; First posted 2014-05-23 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Arthritis of the Knee
Keywords: Arthroplasty, Replacement, Knee/methods; Knee Joint/physiopathology; Knee Joint/radiography; Knee Joint/surgery; Knee Prosthesis; Outcome Assessment (Health Care); Female; Male; Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mechanical alignment (Active Comparator): Patients in this arm will have the Unity Total Knee Replacement System implanted using a surgical technique that utilizes mechanical alignment via measured resection to establish knee alignment.
  Interventions: Device: Unity Total Knee Replacement System
- Anatomic alignment (Active Comparator): Patients in this arm will have the Unity Total Knee Replacement System implanted using a surgical technique that utilizes anatomic alignment via ligament balancing with the tibial cut perpendicular to the tibial anatomic axis.
  Interventions: Device: Unity Total Knee Replacement System

INTERVENTIONS:
Device: Unity Total Knee Replacement System
  Other Names: Unity Total Knee Replacement System (Cruciate Retaining); Unity Total Knee Replacement System (Posterior Stabilised)
  Arms: Mechanical alignment
Device: Unity Total Knee Replacement System
  Other Names: Unity Total Knee Replacement System (Cruciate Retaining); Unity Total Knee Replacement System (Posterior Stabilised)
  Arms: Anatomic alignment

SUMMARY:
This study will compare two different surgical methods used in total knee replacement with the Unity Total Knee Replacement System. The study will evaluate these two methods based on patients' ability to perform various tasks prior to surgery and at 4 time points during the first 12 months after surgery.

DETAILED DESCRIPTION:
This study will be conducted at a single centre. The study has two treatment groups. One group of 50 knees (approximately 50 subjects) will have a surgical method that uses mechanical alignment (alignment based on how the leg and knee joint move) to determine the proper position of the knee replacement device. The other group of 50 knees (approximately 50 subjects) will have a surgical method that uses anatomical alignment (alignment based on how the anatomy/structure of the leg and knee joint) determine the proper position of the knee replacement device. Subjects will be randomly assigned to one of the two groups. Clinical and functional tests will be conducted pre-operatively and at 6 weeks, 3 months, 6 months and 12 months to determine overall knee function. In addition, a CT scan will be completed pre-operatively and at 6 weeks to assess changes in alignment.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be listed for a primary total knee replacement using the Corin Unity Total Knee Replacement System, according to the product 'Instructions For Use'
* The patient must give signed informed consent to participate in the study
* The patient must be able to understand all that is expected of them and be able to comply with the study protocol
* Male and female patients who are skeletally mature

Exclusion Criteria:

* Any patient with a total knee replacement not implanted with a Corin Unity Total Knee Replacement
* Any patient with a revision total knee replacement or conversion of a Unicondylar replacement to a total knee replacement on the operative knee
* Any patient with fixed flexion contracture greater than 20 degrees
* Any patient with varus/valgus deformity greater than 15 degrees
* Any case not described in the inclusion criteria
* Any patient who cannot or will not provide signed informed consent for participation in the study
* Any patient whose prospects for a recovery to independent mobility would be compromised by known co-existent, medical problems
* Any patient with a known sensitivity to device material
* Any patient who is pregnant
* Any patient currently a prisoner
* Any patient known to be a drug or alcohol abuser, or have a psychological disorder that could affect follow-up care or treatment outcomes
* Any patient currently involved in any personal injury litigation, medical-legal or worker's compensations claims
* Any patient unable to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-06-06 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Power of knee extension | 12 months post-operative
  Power of knee extension via peak torque of quads measured on a digital myometer.

SECONDARY OUTCOMES:
Timed up and go test | 12 months post-operative
  The test measures the length of time it takes the subject to rise from a chair, walk 10 feet, turn around, and sit back down in the chair. The subject may rest or use walking aids during the test.
Single leg stance (SLS) test | 12 months post-operative
  The test measures the length of time the subject can stand on their operative leg.
6 minute walk test | 12 months post-operative
  The test measures the length of distance a subject can walk in 6 minutes at a pace that does not cause them to become short of breath. Patient may stop and rest if needed, then resume.
Timed stairs test | 12 months post-operative
  The test measures the length of time it takes a subject to climb up a stair block and down the other side. The subject is asked how difficult the test was on a scale of 0 to 10. The subject can use the rails, if needed.
Wii Fit balance test | 12 months post-operative
  The subject is asked to stand on a Wii Fit balance board while the "Deep breathing" exercise in the Yoga section is selected. The subject is instructed to follow the instructions on the screen. The subject's score is recorded and the subject is asked how difficult the test was on a scale from 1 to 10.
Ability to kneel | 12 months post-operative
  The subject is asked to kneel on a mat on the floor and then rise to a standing position. The subject may use a bench or the floor for balance. After the test, the subject is asked how difficult the test was on a scale of 1 to 10. The subject is allowed to refuse to do the test if he/she feels unable to do so.
Sloped treadmill test | 12 months post-operative
  The subject is asked to walk on a level treadmill at a comfortable walking speed. The incline of the treadmill is increased until the subject says stop or the limit of the treadmill is reached. The test is repeated with the treadmill in reverse and the subject facing backwards to simulate walking downhill. The subject is asked how difficult the test was on a scale of 1 to 10.
Walking on uneven ground | 12 months post-operative
  The subject is asked to walk from one end to the other on a specialized track topped with fist-sized pebbles. The subject is allowed to use walking aids. The subject is asked how difficult the test was on a scale of 1 to 10.
CT evaluation | 6 weeks post-operative
  CT scan will be done to assess the following anatomical items:
  * Medial joint line position
  * Overall limb alignment
  * Joint obliquity
  * Rotation
Power of knee flexion | 12 months post-operative
  Power of knee flexion via peak torque of quads measured on a digital myometer.
Oxford Knee Score (OKS) | 12 months Post-operative
  A questionnaire about your ability to perform daily functions.
Knee Injury and Osteoarthritis Score (KOOS) | 12 months Post-operative
  A questionnaire to assess your ability to perform activities of different difficulty levels.
EuroQoL 5-dimension Health State (EQ-5D) | 12 months Post-operative
  A questionnaire to assess your health and well-being.
Patient Satisfaction Score | 12 months Post-operative
  A questionnaire to assess your satisfaction with your knee implant.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Toms, MD, Principal Investigator — Princess Elizabeth Orthopaedic Centre
Locations (1):
- Exeter Knee Reconstruction Unit at the Princess Elizabeth Orthopaedic Centre, Exeter, Devon, United Kingdom